CLINICAL TRIAL: NCT00136656
Title: Treatment of Acute Pyelonephritis With Gram Negative Strains in Infants and Children Less Than 3 Years Old. Cefixime PO 10d vs Ceftriaxone IV 4d Followed by Cefixime PO 6d. Multicenter, Randomised Trial of Equivalence.
Brief Title: Treatment of Acute Pyelonephritis With Gram Negative Strains in Infants and Children Less Than 3 Years Old
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Thérèse NGOUE, Department Clinical Research of Developpement
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P040422; AOM 04 105
Record Dates: First submitted 2005-08-26; First posted 2005-08-29 (Estimated); Last update posted 2009-02-12 (Estimated); Status verified 2009-02

CONDITIONS: Pyelonephritis
Keywords: infant; children; pyelonephritis; Renal scars; DMSA scan
MeSH Terms: conditions — Pyelonephritis | interventions — Anti-Bacterial Agents

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): cefixime antibiotic treatment by oral route
  Interventions: Drug: antibiotic
- 2 (Sham Comparator): ceftriaxone antibiotic treatment by venous infusion and cefixime antibiotic treatment by oral route during six days
  Interventions: Drug: antibiotics

INTERVENTIONS:
Drug: antibiotic — cephalosporine by oral route : cefixime
  Arms: 1
Drug: antibiotics — cephalosporine : ceftriaxone by intra venous route and cefixime by oral route
  Arms: 2

SUMMARY:
The purpose of this study is to demonstrate the equivalence of the therapeutic efficacy of cefixime by mouth (PO) 10 days (d) and ceftriaxone intravenous route(IV) 4d followed by cefixime PO 6d on renal scars 6 months after a first acute pyelonephritis episode.

The investigators hypothesize that treatment with cefixime PO will allow no more renal scars than intravenous route (IV) treatment of pyelonephritis in infants and children less than 3 years old, 6 months after the first episode. If it is true, treatment will no longer need hospitalisation and the advantages for children, families and the health system will be very important.

DETAILED DESCRIPTION:
Guidelines for treatment of acute pyelonephritis in infants and children are different from one country to another. The main question is the incidence of renal scars.

intravenous route (IV) treatment is supposed to give the best results, but no previous study has ever given the incidence of renal scars after PO treatment.

This multicenter, randomised trial is an equivalence study of PO and intravenous route (IV) treatments.

ELIGIBILITY:
Inclusion Criteria:

* Infants and children more than 1 month old and less than 3 years old
* First episode of acute pyelonephritis with gram negative strains
* Fever more than 38.5°C
* Procalcitonin (PCT) value > 0.5 ng/ml
* Urine obtained by transurethral bladder catheterization, suprapubic aspiration or midstream collection
* Urine exam: more than 100.000 leukocytes and gram negative strains +
* Normal hemodynamic exam
* Normal renal ultrasonography
* Positive DMSA renal scan for pyelonephritis during the first week after diagnosis
* Parental informed consent

Exclusion Criteria:

* Newborn
* Children more than 3 years old
* Past urine infection
* Septic hemodynamic abnormalities
* Obstructive uropathy and any renal ultrasonography abnormalities
* Allergy to cefixime or ceftriaxone
* Antibiotic during the five previous days
* Gastrointestinal abnormalities able to interfere with antibiotic intake or absorption
* Absence of parental consent
* Social familial difficulties

Ages: 1 Month to 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 700 (Actual)
Dates: Start 2005-07; Primary Completion 2008-06 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Renal scars on dimercaptosuccinic acid (DMSA) renal scan at 6 months | between six and eight months

SECONDARY OUTCOMES:
Time to get apyrexia | 4 days
Incidence of urologic abnormalities on cystourethrography done during the first month after the infection | one month

CONTACTS AND LOCATIONS:
Overall Officials: CHERON GERARD, MD, Principal Investigator — Hôpital Necker Enfants Malades Assistance Publique Hôpitaux de Paris - René Descartes University Paris 5; CHEVALLIER BERTRAND, MD, Study Chair — Ambroise Paré Hospital, Assistance Publique Hôpitaux de Paris; GAJDOS VINCENT, MD, Study Chair — Antoine Béclère Hospital Assistance Publique Hôpitaux de Paris; LABRUNE PHILIPPE, MD, Study Chair — Antoine Béclère Hospital Assistance Publique Hôpitaux de Paris; GRIMPREL EMMANUEL, MD, Study Chair — Trousseau Hospital AP HP; DESCHENES GEORGES, MD, Study Chair — TROUSSEAU HOSPITAL AP-HP; SERGENT ALINE, MD, Study Chair — TROUSSEAU HOSPITAL AP-HP; VAYLET CLAIRE, MD, Study Chair — TROUSSEAU HOSPITAL AP-HP; BADER MEUNIER BRIGITTE, MD, Study Chair — BICETRE HOSPITAL AP-HP; GUIGONIS VINCENT, MD, Study Chair — DUPUYTREN HOSPITAL CHU LIMOGES
Locations (12):
- France (12):
  - Hopital de Bicetre, Bicêtre
  - Hopital Pellegrin, Bordeaux
  - Hôpital Ambroise Pare, Boulogne
  - Hôpital Antoine Beclere, Clamart
  - Chu de Limoges, Limoges
  - La Timone, Marseille
  - CHU NICE, Nice
  - Saint Vincent de Paul, Paris
  - Necker Enfants Malades, Paris
  - Robert Debre, Paris
  - Hôpital Armand Trousseau, Paris
  - Hopital Andre Mignot, Versailles

REFERENCES:
- [Background] Sannier N, Le Masne A, Sayegh N, Gaillard JL, Cheron G. Ambulatory management of acute pyelonephritis in children. Acta Paediatr. 2000 Mar;89(3):372-3. No abstract available. PMID 10772296
- [Background] Leroy S, Marc E, Adamsbaum C, Gendrel D, Breart G, Chalumeau M. Prediction of vesicoureteral reflux after a first febrile urinary tract infection in children: validation of a clinical decision rule. Arch Dis Child. 2006 Mar;91(3):241-4. doi: 10.1136/adc.2004.068205. Epub 2005 May 12. PMID 15890693
- [Background] Leroy S, Adamsbaum C, Marc E, Moulin F, Raymond J, Gendrel D, Breart G, Chalumeau M. Procalcitonin as a predictor of vesicoureteral reflux in children with a first febrile urinary tract infection. Pediatrics. 2005 Jun;115(6):e706-9. doi: 10.1542/peds.2004-1631. Epub 2005 May 2. PMID 15867014
- [Background] Marc E, Menager C, Moulin F, Stos B, Chalumeau M, Guerin S, Lebon P, Brunet F, Raymond J, Gendrel D. [Procalcitonin and viral meningitis: reduction of unnecessary antibiotics by measurement during an outbreak]. Arch Pediatr. 2002 Apr;9(4):358-64. doi: 10.1016/s0929-693x(01)00793-x. French. PMID 11998420
- [Derived] Bocquet N, Sergent Alaoui A, Jais JP, Gajdos V, Guigonis V, Lacour B, Cheron G. Randomized trial of oral versus sequential IV/oral antibiotic for acute pyelonephritis in children. Pediatrics. 2012 Feb;129(2):e269-75. doi: 10.1542/peds.2011-0814. Epub 2012 Jan 30. PMID 22291112